CLINICAL TRIAL: NCT03931278
Title: Investigating Auditory Sonification (Melodic and Single Tones) and Visual Real-time Feedback as a Tool for Embodied Associations, and Its Effects on Learning and Balance in Persons With Multiple Sclerosis
Brief Title: Sonification Embodied Associations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Collaborators: University Ghent (Other); Revalidatie & MS Centrum Overpelt (Other); National MS Center Melsbroek (Other)
Responsible Party: Principal Investigator, Peter Feys, Principal Investigator, Hasselt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: SEA-001
Record Dates: First submitted 2019-04-25; First posted 2019-04-30 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- persons with Multiple Sclerosis (MS) (Other)
  Interventions: Other: learning and recall of a sequence of body movements
- Healthy controls (Other)
  Interventions: Other: learning and recall of a sequence of body movements

INTERVENTIONS:
Other: learning and recall of a sequence of body movements — The objective of this study to investigate, if learning and recall of a sequence of body movements (steps that realize a pattern on the ground) can be improved by self-produced music (having particular melodic-structures in relation to the pattern), compared to the same sound (a single tone) for each pattern in persons

SUMMARY:
The objective of this study to investigate, if learning and recall of a sequence of body movements (steps that realize a pattern on the ground) can be improved by self-produced music (having particular melodic-structures in relation to the pattern), compared to the same sound (a single tone) for each pattern in persons with multiple sclerosis compared to age and gender matched controls

ELIGIBILITY:
Inclusion Criteria:

* Time up and Go (TUG) test: 8 sec -- > 21 sec

Exclusion Criteria:

* cognitive impairment hindering the understanding and execution of the experimental procedures,
* pregnancy,
* hearing impairment,
* amusia
* beat deafness,
* colour blindness.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2020-01-24 (Actual); Study Completion 2020-01-24 (Actual)

PRIMARY OUTCOMES:
accuracy | week 1
  Number of correct sequences uttered, total number of sequences, precisions prior to completing three correct trials.
precision | week 1
  Number of correct sequences uttered, total number of sequences, precisions prior to completing three correct trials.

SECONDARY OUTCOMES:
Inter Step intervals | week 1
  The technology used can log time data. Therefore, the inter-step intervals can be calculated from the logged data.
Inter Stride intervals | week 1
  The technology used can log time data. Therefore, the inter stride intervals can be calculated from the logged data.
step duration on the tile | week 1
  The technology used can log time data. Therefore, the total time that each foot is placed on the tiles can be derived.

CONTACTS AND LOCATIONS:
Overall Officials: peter Feys, prof. dr., Principal Investigator — Hasselt University; lousin Moumdjian, Study Chair — Hasselt University
Locations (3):
- Belgium (3):
  - University Ghent, Ghent
  - National MS Center Melsbroek, Melsbroek
  - Revalidatie en MS Centrum Overpelt, Overpelt

IPD SHARING:
Plan to Share IPD: Undecided